CLINICAL TRIAL: NCT03548376
Title: Effects of Hippotherapy in Postural Control, Balance, Gross-motor Function and Quality of Life of Children With Cerebral Palsy
Brief Title: Hippotherapy in Children With Cerebral Palsy
Acronym: Hippotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Marisa Cotta Mancini, Principal Investigator, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMancini
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Cerebral Palsy
Keywords: rehabilitation; cerebral palsy; postural control; balance; gross-motor function; quality of life; hippotherapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Before-after trial (6 months of follow-up; one group with three repeated measurements)
Masking Description: the scoring of repeated evaluations was blinded regarding order. To do so, the scores of all of the instruments were calculated without the knowledge of which was the evaluation (T1, T2 or T3) or access to the previous scores of the same child. The GMFM-88 score was made by an examiner who did not participate in the data collection (evaluations and intervention). This examiner watched the videos and was blinded to the child's descriptive information and the order of the evaluation. The ECAB test score was calculated by two other external examiners who watched the videos and were also blinded regarding the same information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One-group intervention (Experimental): Hippotherapy sessions were delivered once a week for 30 minutes, during 6 months.
  Interventions: Other: Hippotherapy

INTERVENTIONS:
Other: Hippotherapy — Hippotherapy is a therapeutic intervention that is typically conducted by a physical or occupational therapist and is aimed at improving impaired body function. Hippotherapy has been proposed as a technique to decrease the energy requirements and improve walking in patients with cerebral palsy. It is thought that the natural swaying motion of the horse induces a pelvic movement in the rider that simulates human ambulation. In addition, variations in the horse's movements can also prompt natural equilibrium movements in the rider.
  Other Names: horse therapy; equine movement therapy

SUMMARY:
The hippotherapy is a complementary therapeutic modality that seeks to promote changes in the functionality of children with cerebral palsy (CP). Knowing the domains in which this therapy causes both direct and indirect effects, and identify the mechanisms that produce their effects, contributes to broadening and deepening of the knowledge available on the hippotherapy. The main aim of this study was to evaluate changes in postural control and balance, gross motor function and quality of life (QoL) of children with CP undergoing hippotherapy for a period of six months.

DETAILED DESCRIPTION:
We conducted a quasi-experimental study with 31 children with cerebral palsy from both sexes, of various types and GMFCS levels who were followed for 6 months with three repeated measurements: beginning of the study (T1), 3 months (T2) and 6 months (T3) after the initial evaluation. Participants were measured 3 times on postural control and balance, gross-motor function and twice on quality of life. Children attended hippotherapy session one a week for 30 minutes. Sessions were conducted by equestrian therapists (physiotherapists or occupational therapists) qualified by the National (Brazilian) Association of Hippotherapy. The horses were trained for hippotherapy practice, and each patient used the same animal in all sessions. The specific hippotherapy gear included safety straps, riding blankets, stirrups and saddles with and without support straps. The use of protective helmets for patients was mandatory in all sessions. Playful and educational toys were also used. The participants included the patient, the equestrian therapist, the horse handler (the professional who drives the horse) and, when necessary, an auxiliary helper to ensure the safety of the child. The hippotherapy sessions were individualized. The goals set by the therapist were based on the specific demands and the motor condition of each client. The activities proposed during each session sought to stimulate the development of the postural control of the child with CP. Such activities could be performed in various postures (i.e., classic, inverted, lateral, dorsal decubitus, ventral decubitus and standing on the stirrups). They included demands for stability and balance (i.e., trunk rotation activities, range in various directions and bimanual tasks), active stretches and antigravitational exercises during riding, integrated with ludic-cognitive resources (i.e., memory games and identification of colors, numbers and letters). For the most part, children with mild and moderate impairments rode individually and were encouraged to maintain an upright posture throughout the session. Those with more severe impairment were encouraged to maintain control and postural alignment, with the minimum of support being provided. In some cases, it was necessary to use a double riding strategy, in which the therapist rode the horse along with the patient to favor and stimulate the child's postural control on the animal. Throughout the session, the horse varied speed, cadence and direction to the therapist's command, using different paths (i.e., circles, zigzags and straight lines) and different types of terrain (i.e., uphill, downhill, dirt, asphalt and grass). All participants were instructed to continue with their rehabilitation routine (i.e., physical therapy, occupational therapy and others). For data analysis, participants were stratified by age (04-07 years and 08-12 years), severity (mild, moderate and severe), topography of the members involved (diplegia, hemiplegia, and quadriplegia) and previous time of hippotherapy (between 3-6 months and more than 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Children with medical diagnosis of cerebral palsy
* Ages 4 to 12 years old

Exclusion Criteria:

• Other CP-associated diagnoses (e.g., autism)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Child's Postural control and balance | From Pre-intervention to 3 months after intervention onset
  The Early Clinical Assessment of Balance (ECAB) estimates the postural stability of the child according to head and trunk controls during static activities and dynamic activities
Change in Child's Postural control and balance | From 3 months to 6 months after intervention onset
  The Early Clinical Assessment of Balance (ECAB) estimates the postural stability of the child according to head and trunk controls during static activities and dynamic activities

SECONDARY OUTCOMES:
Change in Child's Gross Motor Function Measure (GMFM) | From pre-intervention to 3 months after intervention onset
  Assessed by the GMFM-88, which includes five dimensions: (A) Lying and Rolling, (B) Sitting, (C) Crawling and Kneeling, (D) Standing and (E) Walking, Running and Jumping. The item scores generate a score for each dimension and a total score. Higher scores give information on a greater repertoire of the gross motor function.
Change in Child's Gross Motor Function Measure (GMFM) | From 3 months to 6 months after intervention onset (end on intervention period)
  Assessed by the GMFM-88, which includes five dimensions: (A) Lying and Rolling, (B) Sitting, (C) Crawling and Kneeling, (D) Standing and (E) Walking, Running and Jumping. The item scores generate a score for each dimension and a total score. Higher scores give information on a greater repertoire of the gross motor function.
Change in Child's Quality of Life | From pre-intervention to 6 months after intervention onset (end on intervention period)
  Assessed by the Quality of Life Questionnaire for Children with Cerebral Palsy: questionnaire for primary caregivers (CPQOL-Child), which gives information on the wellbeing of children with CP between 4 and 12 years of age and was administered in an interview with key caregivers. This version has 66 questions organized in seven domains of QOL: social wellbeing and acceptance; functioning; participation and physical health; emotional wellbeing and self-esteem; access to services; pain and disability impact; and family health. Scoring is transformed into domain-specific percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa C Mancini, PhD, Principal Investigator — Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Zadnikar M, Kastrin A. Effects of hippotherapy and therapeutic horseback riding on postural control or balance in children with cerebral palsy: a meta-analysis. Dev Med Child Neurol. 2011;53: 684-691. 2. Whalen CN, Case-Smith J. Therapeutic effects if horseback riding on gross motor function in children with cerebral palsy: a systematic review. Phys Occup Ther Pediatr. 2012;32: 229-242. 3. Meregliano G. Hippotherapy. Phys Med Rehabil Clin North Am. 2004;15: 843-854. 4. Debuse D, Gibb C, Chandler C. Effects of hippotherapy on people with cerebral palsy from the users' perspective: a qualitative study. Phys Theor Pract. 2009;25(3): 174-192.. 5. Davis E, Davies B, Wolfe R, Raadsveld R, Heine B, Thomason P, et al. A randomized controlled trial of the impact of therapeutic horse riding on the quality of life, health, and function of children with cerebral palsy. Dev Med Child Neurol. 2009;51: 111-119. 6. McCoy SW, Bartlett DJ, Yocum A, Jeffries L, Fiss AL, Chiarello L, et al. Development and validity of the early assessment of balance for young children with cerebral palsy. Dev Neurorehabil. 2014; 17: 375-383. 7. Randall KE, Bartlett DK, McCoy SW. Measuring postural stability in young children with cerebral palsy: a comparison of 2 instruments. Pediatr Phys Ther, 2014;26: 332-337. 8. Cyrillo LT, Galvão MCS. Gross Motor Function Measure [GMFM-66 & GMFM-88] (Portuguese translated manual). São Paulo: Memnon; 2011. 9. Russel DJ, Rosenbaum PL, Cadman DT, Gowland C, Hardy S, Jarvis S. The gross motor function measure: a means to evaluate the effects of physical therapy. Dev Med Child Neurol. 1989; 31: 341-352. 10. Russel DJ, Avery LM, Rosenbaum PL, Raina, PS, Walter SD, Palisano RJ. Improved scaling of the gross motor function measure for children with cerebral palsy: evidence of reliability and validity. Physical Therapy, 2000;80: 873-885. 11. Waters E, Maher E, Salmon L, Reddihpugh D, Boyd R. Developing a new quality of life scale for children with cerebral palsy. Child: Care, Health and Develop. 2005; 31: 127-135. 12. Braccialli LMP, Braccialli AC, Sankako AN, Dechandt MLC, Almeida VC, Carvalho SMR. Quality of life questionnaire for children with cerebral palsy (CP QOL-CHILD): Translation and cultural adaptation to the Brazilian Portuguese language. J Hum Growth and Develop. 2013; 23(2): 154-163. 13. Shurtleff TL, Standeven JW, Engsberg JR. Changes in dynamic trunk/head stability and functional reach after hippotherapy. Arch Phys Med Rehabil. 2009;90: 1185-1195. 14. Casady RL, Nichols-Larsen DS. The effect of hippotherapy on ten children with cerebral palsy. Pediatr Phys Ther. 2004;16: 165-172. 15. Park ES, Rha DW, Shin JS, Kim S, Jung S. Effects of hippotherapy on gross motor function and functional performance of children with cerebral palsy. Yonsei Med J. 2014;55(6): 1736-1742. 16. Hammil D, Washington K, White OR. The effect of hippotherapy on postural control in sitting for children with cerebral palsy. Phys Occup Ther Pediatr. 2007;27: 23-42. 17. Galloux P, Richard N, Dronka T, Leard M, Perrot A, Jouffroy JL, et al. Analysis of equine gait using three-dimensional accelerometers fixed on the saddle. Equine Vet J. 1994; 17(Suppl.): 44-47. 18. Temcharoensuk P, Lekskulchai R, Akamanon C, Ritruechai P, Sutcharitpongsa S. Effect of horseback riding simulator on sitting ability of children with cerebral palsy: a randomized controlled trial. J Phys Ther Sci. 2015;27: 273-277.